CLINICAL TRIAL: NCT03958890
Title: A Randomized, Double-blind, Multicenter, Phase III Clinical Trial Comparing HLX10 (Recombinant Anti-pd-1 Humanized Monoclonal Antibody Injection) With Placebo Combined With Chemotherapy (Cisplatin + 5-fu) in the First-line Treatment of Locally Advanced/Metastatic Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: A Clinical Trial Comparing HLX10 With Placebo Combined With Chemotherapy (Cisplatin + 5-fu) in the First-line Treatment of Locally Advanced/Metastatic Esophageal Squamous Cell Carcinoma (ESCC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX10-007-EC301
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLX10 (Experimental)
  Interventions: Drug: HLX10 100 mg in 10 ml Injection
- placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: HLX10 100 mg in 10 ml Injection — 3mg/kg IV（HLX10+cis-platinum+5FU）
  Arms: HLX10
Drug: Placebos — 3mg/kg IV（placebo+cis-platinum+5FU）
  Arms: placebo

SUMMARY:
This study is a randomized, double-blind, multi-center, phase III clinical study comparing the clinical efficacy and safety of HLX10 or placebo combined with chemotherapy in first-line treatment of locally advanced/metastatic esophageal squamous cell carcinoma (ESCC) patients.This study consists of three periods, screening period (28 days), treatment period and follow-up period (including safety follow-up, survival follow-up).Subjects can be enrolled into this study only if they meet inclusion criteria and do not meet exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria are allowed to be enrolled into this study:

  * Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF); be willing to follow and be able to complete all study procedures;
  * Age ≥ 18 years and ≤ 75 years when ICF is signed;
  * Never received systemic anti-tumor drug therapy before.Exception: for patients who have received neoadjuvant/adjuvant treatment, the time from the last treatment to recurrence or progression can be screened for more than 6 months;For patients who have received radical concurrent chemoradiotherapy or radiotherapy for esophageal cancer, the time from the last chemotherapy/radiotherapy to the recurrence or progression time is more than 12 months.
  * According to the curative effect evaluation criteria in solid tumors (RECIST) v1.1, assessed by the center image with at least one measurable lesions (such as esophageal cavity structure not as measurable lesions), measurable lesions should be not received radiotherapy, etc (lesions located in the usual radiation area, if confirm progress, can also be selected as the target lesion);
  * PD-L1 positive subjects (CPS 1%).The subject must provide tumor tissue for pd-l1 expression level determination;
  * Within 7 days before the first use of the study drug, ECOG: 0 ~ 1;
  * Expected survival 12 weeks;
  * The functions of the vital organs meet the following requirements (no blood transfusion, cytokine growth factor, or platelet raising drugs are allowed within 14 days before the first use of the study drugs); H. Absolute neutrophil count (ANC) ≥1.5 109/L I. platelet≥ 100 109/L; J. Hemoglobin≥ 9g/dL; K. Serum albumin≥ 3.0g/dL; L. Total bilirubin≤ 1.5 ULN, ALT, AST and/or ALP≤ 2.5 ULN;ALT and/or AST≤ 5 ULN in the presence of liver metastasis;If there is liver metastasis or bone metastasis ALP≤ 5 ULN; M. Serum creatinine ≤1.5 ULN or creatinine clearance > 60 mL/min (Cockcroft-Gault formula); N. APTT, INR and PT ≤1.5 ULN;
  * For fertile female subjects, the serum pregnancy test must be negative within 7 days before the first dose.With fertile women subjects, and the partner for childbearing age women of male subjects, needs during the therapy, and after the last use HLX10 / placebo at least 3 months and the last time to use at least 6 months after chemotherapy using an approved by the medical contraception (such as intrauterine device, the pill or condoms);
  * Subjects voluntarily participated in this study and signed the informed consent, with good compliance and follow-up.

Exclusion Criteria:

* Subjects who meet any of the following criteria are not allowed to be enrolled in this study:

  * 1. BMI < 17.5kg /m2;
  * 2. A history of gastrointestinal perforation and/or fistula within 6 months prior to the first administration;
  * 3. Obvious invasion of tumor into adjacent organs (aorta or trachea) of esophageal lesions leads to high risk of bleeding or fistula;3. Subjects after endotracheal stent implantation;
  * 4. Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage;
  * 5. Previous allergies to monoclonal antibody, HLX10, 5-fu, cisplatin and other platinum drugs;
  * 6.Have received any of the following treatments: A. Previous treatment with anti-pd-1 or anti-pd-L1 antibodies; B. Have received any research drugs within 4 weeks before the first use of the study drugs; C. Be enrolled in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or a follow-up interventional clinical study; D. Receive the final anticancer treatment within 4 weeks before the first use of the study drug;Palliative radiotherapy for bone metastases was allowed and was completed 2 weeks before the first dose.Radiotherapy covering more than 30% of the bone marrow area is not allowed within 28 days before the first dose.

E. Subjects who require systemic treatment with corticosteroids (> 10 mg/ day prednisone therapeutic dose) or other immunosuppressive agents within 14 days prior to the first use of the study drug;In the absence of active autoimmune disease, inhalation or topical use of steroids is permitted, and the therapeutic dose of prednisone 10mg/ day is allowed.

F. Those who have received the anti-tumor vaccine or the live vaccine within 4 weeks before the first dose of the study drug; G. Have undergone major surgery within 28 days prior to the first use of the study drug. Major surgery in this study is defined as requiring at least 3 weeks of postoperative recovery time before being able to receive the surgery treated in this study.Tumor puncture or lymph node biopsy were allowed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years
  Progression-free survival (assessed by independent radiological review committee (IRRC) based on RECIST v1.1)
OS | from the date of first dose unitl the date of death from any cause，assessed up to 2 years
  Overall survival (OS)

SECONDARY OUTCOMES:
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years
  Progression-free survival (assessed by independent radiological review committee (IRRC) based on iRECIST，by the investigators based on RECIST v1.1))
ORR | up to 2 years
  Objective response rate (assessed by independent radiological review and the investigators based on RECIST v1.1))
Duration of response | from the date when CR or PR (whichever recorded earlier) is firstly achieved until the date when disease progression or death is firstly recorded (whichever occurs earlier),assessed up to 2 years
  Duration of response

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Ethics Committeeof cancer hospital, Chinese academy of medical sciences,, Beijing, Beijing Municipality
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Affiliated Tumor Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The first Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - the affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - the second Hospital of Jilin University, Changchun, Jilin

REFERENCES:
- [Derived] Liu S, Jiang N, Dou L, Li S. Cost-effectiveness analysis of serplulimab plus chemotherapy in the first-line treatment for PD-L1-positive esophageal squamous cell carcinoma in China. Front Immunol. 2023 May 4;14:1172242. doi: 10.3389/fimmu.2023.1172242. eCollection 2023. PMID 37215110
- [Derived] Song Y, Zhang B, Xin D, Kou X, Tan Z, Zhang S, Sun M, Zhou J, Fan M, Zhang M, Song Y, Li S, Yuan Y, Zhuang W, Zhang J, Zhang L, Jiang H, Gu K, Ye H, Ke Y, Li J, Wang Q, Zhu J, Huang J; ASTRUM-007 investigators. First-line serplulimab or placebo plus chemotherapy in PD-L1-positive esophageal squamous cell carcinoma: a randomized, double-blind phase 3 trial. Nat Med. 2023 Feb;29(2):473-482. doi: 10.1038/s41591-022-02179-2. Epub 2023 Feb 2. PMID 36732627
- See also: First-line serplulimab or placebo plus chemotherapy in PD-L1-positive esophageal squamous cell carcinoma: a randomized, double-blind phase 3 trial — https://doi.org/10.1038/s41591-022-02179-2
- See also: First-line serplulimab versus placebo in combination with chemotherapy in PD-L1-positive oesophageal squamous cell carcinoma (ASTRUM-007): A randomised, double-blind, multicentre phase III study — https://doi.org/10.1016/j.annonc.2022.10.105